CLINICAL TRIAL: NCT03724097
Title: Identification of Molecular Biomarkers for Cancer Target Therapy Efficacy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OmicsWay Corp. (Industry)
Collaborators: Oncobox Ltd (Unknown); Vitamed LLC (Unknown); N.N. Blokhin National Medical Research Center of Oncology (Other); Kaluga Regional Clinical Oncology Center (Other); Multidisciplinary medical holding SM-Clinic (Unknown); Oncological Clinical Dispensary No. 1 of the Moscow City Health Department (Unknown)
Responsible Party: Sponsor
Other Study IDs: OB0052018
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Cancer
Keywords: biomarkers; target therapy; NGS; RNAseq; mRNA; transcriptome analysis; signaling pathway; intracellular molecular pathway; Oncobox; Next generation sequencing; RNA sequencing
MeSH Terms: conditions — Neoplasms | interventions — Sequence Analysis, RNA; RNA-Seq; Gene Expression Profiling; Drug Delivery Systems; Palliative Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Formalin-fixed, paraffin-embedded pathological cancer samples obtained during surgery or core needle biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Group 1: Patients receiving target drugs with the score value above 0,1 as monotherapy or in combination
  Interventions: Other: RNA sequencing; Other: Transcriptome analysis; Drug: target drug with the score above 0,1
- Group 2: Patients receiving only non-target drugs or target drugs with the score value equal to or below 0,1 as monotherapy or in combination
  Interventions: Other: RNA sequencing; Other: Transcriptome analysis; Drug: target drug with the score equal or below 0,1; Drug: non-target drug
- Group 3: Patients receiving palliative care
  Interventions: Other: RNA sequencing; Other: Transcriptome analysis; Drug: palliative care

INTERVENTIONS:
Other: RNA sequencing — Next Generation Sequencing of RNA from tumor samples, rRNA-depleted.
  Other Names: RNA-seq
Other: Transcriptome analysis — Analysis of RNA-seq data using the Oncobox algorithm.
Drug: target drug with the score above 0,1 — target drug with the score above 0,1
  Groups: Group 1
Drug: target drug with the score equal or below 0,1 — target drug with the score equal or below 0,1
  Groups: Group 2
Drug: non-target drug — non-target drug
  Groups: Group 2
Drug: palliative care — palliative care
  Groups: Group 3

SUMMARY:
This is a prospective trial for a computation-based efficacy prediction method for anticancer target therapies. The original computational algorithm utilizes individual transcriptome data of a cancer sample and assesses changes at the level of gene expression and intracellular signaling pathways. By applying the database of known molecular targets of anticancer target drugs it allows to rank potential efficacies of target drugs.

DETAILED DESCRIPTION:
Original computational algorithm Oncobox was developed to determine molecular features of individual tumors. It represents the solution for a personalized selection of target anticancer therapies. The method is based on the analysis of gene expression profile of a cancer sample in comparison with the corresponding normal tissue biosamples in order to select the most effective molecular targets for their inhibition and, accordingly, to identify more effective target drugs for cancer treatment. Histological material obtained from cancer patients during surgery or core-needle biopsy as part of standard treatment will be used for the analysis. Total RNA extracted from the tumor material will be subjected to next-generation sequencing (NGS). By comparing transcriptome profile of the tumor sample with the profiles of the corresponding normal tissue samples the rate of molecular pathways activation/deactivation will be calculated, as well as the case-to-normal ratios for the individual gene products - molecular targets of drugs. Based on these data, each target drug will be assigned with a score reflecting its potential efficacy for each individual tumor treatment. A drug with the score value above 0.1 will be considered potentially effective, a drug with the score value equal to or below 0.1 - as potentially ineffective. Following Oncobox test, 130 target anticancer drugs will be rated according to their predicted effectiveness (see the list of eligible target drugs below). This information will be fully available to a patient and his/her doctor. The doctor will prescribe treatment according to his/her consideration, e.g. based on the standards of care and the patient's life indications. After the appointment of therapy, the patients will be divided naturally into the following three observation groups. The first group will be formed from patients receiving target drugs with the score value above 0,1 as monotherapy or in combination. The second group - patients receiving only non-target drugs or target drugs with the score value equal to or below 0,1 as monotherapy or in combination. Third group will be formed by patients receiving palliative care. Within this study, these three groups will be compared by response to the therapy according to the results of instrumental studies, by time to progression and by time to progression compared to the previous line of therapy (if any). Additionally, overall survival will be measured in all three groups.

Eligible target drugs:

1. Abemaciclib (LY2835219)
2. Afatinib
3. Aflibercept
4. Alectinib
5. Alemtuzumab
6. Alitretinoin
7. Anastrozole
8. Apalutamide, ARN-509
9. Arsenic trioxide
10. Atezolizumab
11. Avelumab
12. Axitinib
13. Belinostat
14. Bevacizumab
15. Bexarotene
16. Bicalutamide
17. Binimetinib (MEK162)
18. Blinatumomab
19. Bortezomib
20. Bosutinib
21. Brentuximab vedotin
22. Brigatinib
23. Cabazitaxel
24. Cabozantinib
25. Carfilzomib
26. Ceritinib (Zykadia, LDK378)
27. Cetuximab
28. Cobimetinib
29. Crizotinib
30. CYT387 (Momelotinib)
31. Dabrafenib
32. Daratumumab
33. Dasatinib
34. Degarelix
35. Denileukin diftitox (Ontac)
36. Denosumab
37. Docetaxel
38. Dovitinib
39. Durvalumab
40. Elotuzumab
41. Encorafenib
42. Enzalutamide
43. Erlotinib
44. Estramustine
45. Everolimus
46. Exemestane
47. Flavopiridol (Alvociclib)
48. Foretinib
49. Fulvestrant
50. Ganetespib (STA-9090)
51. Gefitinib
52. Goserelin
53. Homoharringtonine (Omacetaxine mepesuccinate)
54. Ibritumomab tiuxetan
55. Ibrutinib
56. Idelalisib
57. Imatinib
58. Inotuzumab ozogamicin
59. Ipilimumab
60. Ixabepilone
61. Ixazomib (MLN9708)
62. Lapatinib
63. Lenalidomide
64. Lenvatinib
65. Letrozole
66. Leuprolide
67. Lomustine
68. Masitinib
69. Medroxyprogesterone acetate (MPA)
70. Megestrol
71. Methyltestosterone
72. Midostaurin
73. Mogamulizumab
74. Moxetumomab pasudotox
75. Necitumumab
76. Nilotinib
77. Nilutamide
78. Nimotuzumab
79. Nintedanib (BIBF 1120)
80. Niraparib
81. Nivolumab (BMS-936558)
82. Obinutuzumab
83. Ofatumumab
84. Olaparib
85. Olaratumab
86. Osimertinib
87. Paclitaxel
88. Palbociclib
89. Panitumumab
90. Panobinostat
91. Pazopanib
92. Pembrolizumab
93. Perifosine
94. Pertuzumab
95. Pomalidomide
96. Ponatinib
97. Ramucirumab (Cyramza)
98. Regorafenib
99. Ribociclib
100. Rigosertib
101. Rituximab
102. Romidepsin
103. Rucaparib
104. Ruxolitinib
105. Selumetinib
106. Siltuximab
107. Sonidegib (LDE225)
108. Sorafenib
109. Sunitinib
110. Tamoxifen
111. Tecemotide (Emepepimut-S, L-BLP25)
112. Temozolomide
113. Temsirolimus
114. Thalidomide
115. Tivantinib
116. Tivozanib
117. Toremifene
118. Trametinib (Mekinst)
119. Trastuzumab
120. Trebananib
121. Vandetanib
122. Veliparib
123. Vemurafenib
124. Venetoclax
125. Vinblastine
126. Vincristine
127. Vindesine
128. Vinorelbine
129. Vismodegib
130. Vorinostat

ELIGIBILITY:
Inclusion Criteria:

* Adults, diagnosed with cancer;
* Age 18 - 80;
* Patients who previously received anticancer treatment within the standard care, patients for whom standard therapy was not indicated or patients refused to receive standard therapy. Patients could receive an unlimited number of treatment lines before this study;
* Available formalin fixed, paraffin-embedded (FFPE) samples of cancer tissue. The material should be confirmed by a certified pathologist, the sample taken for the analysis should contain at least 70% of tumor cells;
* Anticipated survival of at least 3 months since the patient's inclusion in the current investigation;
* Patients who have signed an informed consent.

Exclusion Criteria:

* Anticipated survival of less than 3 months since the patient's inclusion in the current investigation;
* Lack of tumor biopsy material, inability to obtain a new tumor biopsy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncological patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response | 2 years
  Tumor response according to the results of instrumental studies
Time to progression | 2 years
  Time to progression
Time to progression compared to the previous therapy lane | 2 years
  Time to progression compared to the previous therapy lane

SECONDARY OUTCOMES:
Overall survival | 2 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Anton A Buzdin, Ph.D., D.Sc, Principal Investigator — OmicsWay Corp.
Locations (7):
- OmicsWay Corp., Walnut, California, United States
- Russia (6):
  - Kaluga Regional Clinical Oncology Center, Kaluga
  - Oncological Clinical Dispensary No. 1 of the Moscow City Health Department, Moscow
  - Multidisciplinary medical holding "SM-Clinic", Moscow
  - N.N. Blokhin National Medical Research Center of Oncology, Moscow
  - "Oncobox" Ltd., Moscow
  - Vitamed LLC, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan (SAP), NGS data, Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 3 months after trial completion, no end date
Access Criteria: Anyone